CLINICAL TRIAL: NCT03654820
Title: Effectiveness of Using Silver Diammine Fluoride Solution and Combination of Povidone Iodine and Sodium Fluoride Varnish in Preventing Dental Root Caries in Elders: a Randomized, Double-blind, Non-inferiority Trial
Brief Title: Effectiveness on SDF Solution and PVP-I Combined NaF Varnish in Preventing Root Caries in Elders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW 16-162
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Root Caries
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVP-I solution combined with NaF varnish (Experimental): 4-monthly application of 10% povidone-iodine solution and 5% sodium fluoride varnish
  Interventions: Device: PVP-I solution combined with NaF varnish
- SDF treated (Active Comparator): Annual application of 38% SDF solution
  Interventions: Device: SDF solution

INTERVENTIONS:
Device: PVP-I solution combined with NaF varnish — 4-monthly application of 10% povidone-iodine solution and 5% sodium fluoride varnish
  Arms: PVP-I solution combined with NaF varnish
Device: SDF solution — Annual application of 38% SDF solution
  Arms: SDF treated

SUMMARY:
The main objective of this study is to compare the effectiveness and cost-effectiveness of 4-monthly application of 10% povidone iodine solution followed by 5% sodium fluoride varnish with those of annual application of 38% silver diammine fluoride solution on the prevention of new dental root caries in elders. A secondary objective is to compare the effectiveness of the two interventions mentioned above on arresting (halting the progression) active root surface caries in the elders, thus avoiding the need for placing dental restorations.

This proposed study is a randomized double-blind controlled clinical trial with 24-month follow-up. A total of 353 elders aged 60 years or above living in residential homes or attending long-term care facilities in different districts in Hong Kong were recruited. Baseline clinical examination will be conducted by two calibrated examiners in the homes using an intra-oral LED light, dental mirrors and probes. Subjects were randomly allocated to one of the two study groups:

1) positive control - received annual application of 38% silver diammine fluoride solution; and 2) test - received application of 10% povidone iodine solution followed by application of 5% sodium fluoride varnish every 4 months. Follow-up examinations will be carried out after 12 and 24 months by the same blinded examiners to assess the clinical outcomes, i.e. whether new dental caries has developed and whether the active root surface caries lesions found at baseline have become arrested (hardened).

DETAILED DESCRIPTION:
The study population of this proposed clinical trial is adults aged 60 years and above living in residential care homes or attending long-term care facilities in Hong Kong. Totally, 10 residential care homes or long-term care institutions served by NGO dental outreach teams in various districts with different background were selected by the PI in consultation with the NGOs. All elders living in the selected residential homes were invited to attend a free dental examination. Elders fulfilling the inclusion criteria were invited to participate in this study and informed written consent will be obtained before commencement of the study. Dental treatments other than the study interventions were provided by dentists from the NGOs which serve the residential homes.

Totally, 353 elder adults enrolled in the trial. The baseline examination was carried out in the residential home by two calibrated examiners, and so will be as follow-up examinations after 12 and 24 months. A portable dental chair, an intra-oral LED light, disposable dental mirrors and CPI probes were used in the examination.

For each tooth that was not indicated for extraction, status of its crown and its root were assessed and recorded separately. Caries diagnosis was based on visual and tactile inspection. No radiograph was taken. Plaque and food debris that obscures visual inspection of the tooth surfaces were removed. Four surfaces (mesial, distal, buccal and lingual) per tooth were examined and the status were recorded using the following codes which basically follow the criteria recommended by the International Caries Detection and Assessment System (ICDAS II) Coordinating Committee (2009).

The oral hygiene status of the subject was assessed and recorded by using the Visible Plaque Index (Ainamo & Bay, 1975). The presence or absence of visible plaque were recorded on four surfaces (mesial, distal, buccal and lingual) per tooth.

The gingival status of the subject was assessed and recorded using the Gingival Bleeding Index (Ainamo & Bay, 1975). The presence or absence of bleeding within 10 seconds after running a probe across the gingival margin was recorded on four surfaces (mesial, distal, buccal and lingual) per tooth.

Other information that was recorded included whether the subject normally wears a removable partial denture or not, and the subject's general health status and medications that affect the saliva flow rate.

The same calibrated two examiners were blinded by the assignment of the participants. A random sample of 10% of the subjects were re-examined during each examination to monitor intra-examiner reproducibility.

At the examinations, the subjects were asked to report on their oral hygiene practices, use of fluoridated toothpaste and other topical fluoride agents, and use of dental services during the study period.

Oral health education talk and instructions on how to keep good oral hygiene were provided at baseline and every year to all the elders in the selected residential homes. Standard fluoride toothpastes with 1000-1500 ppm fluoride were provided free to all the elders in the selected residential homes over the 24-month study period.

After the baseline examination, subjects satisfying the inclusion criteria of the study were stratified into two groups according to the number of natural teeth with exposed root surfaces in their mouth, those with 12 or fewer teeth and those with 13 or more teeth. The subjects were assigned to one of the two study groups by a research assistant using a block randomization method with a block size of 6. The stratified randomization procedure will help to ensure that the numbers of teeth involved in the two study groups are balanced. The interventions for the two study groups were provided by other dentists and are described below:

Group 1 - plaque on the root surfaces of all teeth in the subject's mouth was removed and a 38% SDF solution (Saforide, Toyo Chemical, Japan ) was applied onto the root surfaces using a microbrush/applicator. This will be repeated every year.

Group 2 - plaque on the root surfaces of all teeth in the subject's mouth was removed and a 10% povidone iodine solution (Betadine, Mundipharma, Switzerland) was applied, then followed by application of a 5% sodium fluoride varnish (Duraflor, Medicom, Canada) using a microbrush/applicator. This will be repeated every 4 months.

ELIGIBILITY:
Inclusion Criteria:

* have at least 6 teeth which are not indicated for extraction, and
* have basic self-care ability.

Exclusion Criteria:

* have serious debilitating health/medical conditions, and
* have cognitive problems or major problems in communication.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
new root caries found in clinical examination | 24 months
  development of new carious lesion on exposed tooth root as assessed in clinical examination where there is a soft decayed root surface on gentle probing with a blunt probe

SECONDARY OUTCOMES:
arrested root caries found in clinical examination | 24 months
  in the follow-up clinical examination, there is arrest of active caries lesions that were present at baseline and found to be a hard root surface upon gentle probing with a blunt probe

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03654820/Prot_001.pdf